CLINICAL TRIAL: NCT02608723
Title: Chronic Plantar Fasciitis Treated With Shock Wave Therapy: Do the External Appearance of the Device Influence Clinical Outcomes? A Randomized Controlled Clinical Trial.
Brief Title: Shock Wave Therapy: Do the External Appearance of the Device Influence Clinical Outcomes?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asociacion Colaboracion Cochrane Iberoamericana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1304
Record Dates: First submitted 2015-11-13; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Plantar Fasciitis; Pain
Keywords: shock wave; plantar fasciitis; placebo effect; nocebo effect
MeSH Terms: conditions — Fasciitis, Plantar; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard shock waves device (Active Comparator): 3 sessions were applied: one per week.
  Interventions: Device: Standard shock waves device
- Austere shock waves device (Active Comparator): 3 sessions were applied: one per week.
  Interventions: Device: Austere shock waves device
- Sophisticated shock waves device (Active Comparator): 3 sessions were applied: one per week.
  Interventions: Device: Sophisticated shock waves device

INTERVENTIONS:
Device: Standard shock waves device — 3 sessions were applied: one per week. Energy flux density 0,18 mJ/mm2. Frequency: 8 Hz. 2500 shockwaves/session. The shock waves emitted to the 3 devices are identical; the only difference is the external image of the device.
  Arms: Standard shock waves device
Device: Austere shock waves device — 3 sessions were applied: one per week. Energy flux density 0,18 mJ/mm2. Frequency: 8 Hz. 2500 shockwaves/session. The shock waves emitted to the 3 devices are identical; the only difference is the external image of the device.
  Arms: Austere shock waves device
Device: Sophisticated shock waves device — 3 sessions were applied: one per week. Energy flux density 0,18 mJ/mm2. Frequency: 8 Hz. 2500 shockwaves/session. The shock waves emitted to the 3 devices are identical; the only difference is the external image of the device.
  Arms: Sophisticated shock waves device

SUMMARY:
To check in patients suffering from chronic plantar fasciitis treated with shock wave therapy, if the outward appearance of the device affects clinical outcomes.

DETAILED DESCRIPTION:
Study Design: a controlled, randomized, parallel assessor-blinded clinical trial.

Patients suffering from chronic plantar fasciitis (duration more than 6 months) will be assigned to three different groups:

* Group I: Treatment applied by standard shock waves device.
* Group II: Shock wave therapy applied by a modified standard device to offer more attractive, more technical, smarter, better appearance, larger and with an expansion of external information devices more sophisticated.
* Group III: Shock wave therapy applied by a modified standard device to offer a more austere, disfigured, unattractive, modest and smaller external appearance.

The shock waves emitted to the 3 devices will be identical; the only difference will be the external image of the device.

The main outcome will be the function of the foot by the FFI (Foot Function Index) questionnaire.

As secondary variables: pain by VAS (Visual Analogical Scale) in different situations, the plantar fascia thickness measured by ultrasound, and the perception of patient recovery measured with the Likert scale. Adverse effects, painkillers consumption and pain experienced during the treatment of shock waves were also assessed.

The patients will be followed and monitored for a month, two months and four months after treatment finished.

For the statistical analysis of clinical variables, ANOVA (analysis of variance) will be performed to check whether the evolution of patients over time was different depending on the device applied.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years.
2. Being able to understand the explanations about the potential benefits and risks of study participation.
3. Diagnosis of chronic plantar fasciitis. Proven by clinical examination: Meeting at least 2 of the following criteria:

   * Tenderness in the proximal insertion of the plantar fascia (area of the medial calcaneal tuberosity).
   * Pain during the first steps to get out of bed in the morning and / or after a period of rest time.
4. With a duration of symptoms ≥ 6 months at the time of study entry.
5. Having received conservative therapy without success, at least two treatments. Treatments may have been made isolated, combined or consecutively.

Exclusion Criteria:

1. Bilateral plantar fasciitis.
2. Hiper/ hypothyroidism.
3. Diabetes mellitus.
4. Treatment with anticoagulants
5. Inflammatory diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Function of the foot | Four months
  FFI (Foot Function Index) questionnaire

SECONDARY OUTCOMES:
Pain | Four months
  VAS (Visual Analogical Scale)
Plantar fascia thickness | Four months
  Ultrasounds
Perception of patient recovery | Four months
  Likert scale
Painkillers consumption | Four months
  Painkillers consumption
Adverse effects | Four months
  Adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Morral, PhDc, Principal Investigator — Rehabilitation Center "Salut i Esport"
Locations (1):
- Rehabilitation Center "Salut i Esport", Santa Perpètua de Gaià, Barcelona, Spain